CLINICAL TRIAL: NCT00909428
Title: Validation of a Real-time Urodynamic Measure of Urinary Urgency as a Measure of the Success of Drug Treatment
Brief Title: Validation of a Real-time Urodynamic Measure of Urinary Urgency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109248
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Overactive Bladder Syndrome
Keywords: Bladder; Urinary Urgency; Solifenacin; Vesicare(R)
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Solifenacin Succinate (Experimental): The intervention for this study is 10mg daily solifenacin. Patients with overactive bladder syndrome will take this study drug for 30 days.
  Interventions: Drug: Solifenacin Succinate

INTERVENTIONS:
Drug: Solifenacin Succinate — Participants take 10mg daily solifenacin succinate for 30 days
  Other Names: Vesicare(R)

SUMMARY:
Urinary urgency is a key symptom of overactive bladder syndrome (OAB) and may be more bothersome to a patient than the symptom of urinary frequency. Unfortunately, controversy continues to surround the term 'urgency' and there is no good tool to evaluate the severity of urgency. This fact has constrained the performance of clinical research in this field. The cause of urinary urgency is not fully understood and may vary from patient to patient.

Although clinicians regularly obtain measures of bladder sensation during cystometry, little attention has been paid to the patient experience of urinary urgency. In this study, the researchers will use a non-significant risk device (i.e., an Urgeometer) to measure urinary urgency in women with overactive bladder.

DETAILED DESCRIPTION:
At baseline, a small catheter is placed inside the participant's bladder. The bladder is filled with sterile water through the catheter. As the bladder is filled, the participant is asked to rate their urinary urgency using the Urgeometer. The Urgeometer lever marks a continuous scale from 0 'no urge at all' to 100 'maximum urge which you can tolerate'. The testing is stopped once the bladder is filled. To minimize the chance of infection, participants receive one dose of oral antibiotics prior to the bladder testing.

Following completion of the bladder test, participants will take 10mg solifenacin succinate (VesicareR) daily for 30 days. Afterward, participants repeat the bladder test. The change in participants' maximal tolerated cystometric capacity (MCC) will be measured in milliliters and used to evaluate the effectiveness of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Have symptoms of urge or mixed incontinence (urge predominant) and desire treatment with anticholinergic medication.
* Demonstrated detrusor overactivity with or without incontinence during urodynamic testing.
* Are able to consent and fill out study documents, complete repeated urodynamic testing, and follow-up in 4 weeks.

Exclusion Criteria:

* Have been treated with any anticholinergic medication in the previous month.
* Have an elevated post -void residual volume as determined during their routine clinical care.
* Have had a urinary tract infection in the last month, as determined by history.
* Have untreated narrow angle glaucoma, by patient history.
* Have a known allergy or intolerance to solifenacin, as determined by patient history.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary P FitzGerald, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Due to restrictions on the availability of individual participant data (IPD), IPD are not publicly available

REFERENCES:
- [Background] Craggs MD. Objective measurement of bladder sensation: use of a new patient-activated device and response to neuromodulation. BJU Int. 2005 Sep;96 Suppl 1:29-36. doi: 10.1111/j.1464-410X.2005.05649.x. PMID 16086677
- [Background] Oliver S, Fowler C, Mundy A, Craggs M. Measuring the sensations of urge and bladder filling during cystometry in urge incontinence and the effects of neuromodulation. Neurourol Urodyn. 2003;22(1):7-16. doi: 10.1002/nau.10082. PMID 12478595
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Background] Herzog AR, Diokno AC, Fultz NH. Urinary incontinence: medical and psychosocial aspects. Annu Rev Gerontol Geriatr. 1989;9:74-119. doi: 10.1007/978-3-662-40455-3_3. PMID 2514773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-one individuals were consented and 42 women with overactive bladder (OAB) received study drug between January 2007 and February 2009. Participants were recruited using physician solicitation.
Pre-assignment Details: Following informed consent, nine women were negative for OAB and did not receive solifenacin succinate
Groups:
- Detrusor Overactivity Incontinence (DOI): Patients in this cohort were diagnosed with detrusor overactivity incontinence (DOI).
- Urodynamic Stress Incontinence (USI): Patients in this cohort were diagnosed with urodynamic stress incontinence (USI)
- Mixed Incontinence (DOI-USI): Patients in this cohort were diagnosed with both detrusor overactivity incontinence (DOI) and urodynamic stress incontinence (USI)
Period: Overall Study
Arm/Group | Detrusor Overactivity Incontinence (DOI) | Urodynamic Stress Incontinence (USI) | Mixed Incontinence (DOI-USI)
Started | 18 | 15 | 9
Completed | 5 | 5 | 0
Not Completed | 13 | 10 | 9
Not completed — Lost to Follow-up | 13 | 10 | 9

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all women who signed informed consent and have a valid diagnosis of OAB
Groups:
- Total: Total of all reporting groups
Arm/Group | Detrusor Overactivity Incontinence (DOI) | Urodynamic Stress Incontinence (USI) | Mixed Incontinence (DOI-USI) | Total
Number analyzed (Participants) | 18 | 15 | 9 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 9 | 34
  >=65 years | 4 | 4 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 9 | 42
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Cystometric Capacity (mL)
Description: At baseline, a small catheter is placed inside the participant's bladder. The bladder is filled with sterile water through the catheter and participants' maximal tolerated cystometric capacity (MCC) is measured in milliliters. Following completion of the bladder test, participants take 10mg solifenacin succinate (VesicareR) daily for 30 days. After 30 days of treatment, participants repeat the bladder test. Change in the MCC is used to evaluate the effectiveness of the drug.
Time Frame: 30 Days
Population: The primary outcome analysis population comprises only women with two valid MCC recordings (i.e., one baseline recording and one recording following 30 days of treatment with daily 10mg solifenacin succinate. The groups DOI and USI were combined for this repeated measures analysis.
Measure: Median (Inter-Quartile Range); unit: milliliters (mL)
Groups:
- Baseline Maximal Cystometric Capacity: All patients with DOI or USI had their baseline maximal cystometric capacity recorded
- One Month Maximal Cystometric Capacity: All patients with DOI or USI had their maximal cystometric capacity recorded following 30 days of treatment with daily 10mg solifenacin succinate.
Arm/Group | Baseline Maximal Cystometric Capacity | One Month Maximal Cystometric Capacity
Number analyzed (Participants) | 10 | 10
milliliters (mL) | 95 [0 to 99.25] | 473.50 [416.75 to 549.50]
Statistical Analysis 1: Comparison: Baseline Maximal Cystometric Capacity vs One Month Maximal Cystometric Capacity; The null hypothesis is that there is no change from baseline maximal tolerated cystometric capacity following 30 days of treatment with daily 10mg solifenacin succinate; Test type: Superiority; p = .005, Wilcoxon signed rank test; Z-Score = 2.803

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 30 day trial
Arm/Group | Detrusor Overactivity Incontinence (DOI) | Urodynamic Stress Incontinence (USI) | Mixed Incontinence (DOI-USI)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/9

LIMITATIONS AND CAVEATS:
The trial experienced significant attrition. Otherwise, there are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No